CLINICAL TRIAL: NCT06486493
Title: Effectiveness of a Family Playful / Ludic Educational Strategy Reinforced With the Use of Information and Communication Technologies in the Prevention and Reduction of Childhood Obesity
Brief Title: Impact of a Playful Family Education Strategy With ICT on Childhood Obesity Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Doctorado en Ciencias Biomédicas, Universidad Nacional Autónoma de México (Unknown); Facultad de Medicina, Universidad Nacional Autónoma de México (Unknown); Escuela Superior de Medicina, Instituto Politécnico Nacional (Unknown); Instituto Nacional de Salud Pública (Unknown)
Responsible Party: Principal Investigator, José de Jesús Peralta Romero, Principal investigator, head of clinical department of the Unidad de Investigación Médica en Bioquímica, Unidad Médica de Alta Especialidad "Dr. Bernardo Sepúlveda", Centro Médico Nacional Siglo XXI, IMSS, Mexico City, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-2020-785-036; 0594 (Other Grant/Funding Number: Instituto Mexicano del Seguro Social (IMSS)); 09-CEI-009-20160601 (Other: CONBIOÉTICA); 17 CI 09 015 006 (Other: COFEPRIS)
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Obesity; Childhood Obesity; Childhood Overweight
Keywords: Pediatric Obesity; Childhood Obesity; Educational Activities; Technology
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Overweight conventional treatment group (Active Comparator): Children between 9 to 12 years old, from the Family Medicine Unit No. 1 and 3 (IMSS, Morelos) with a BMI Z-score 1 to 2 standard deviations above the median of the established growth patterns by age and sex, and a BMI above the 85th percentile, according to the World Health Organization (WHO) and the Centers for Disease Control and Prevention (CDC). Who will be treated with conventional medical treatment by their physicians, following the Clinical Practice Guideline for the Prevention and Diagnosis of Overweight and Obesity in Children and Adolescents (SS-025-08) and the Guideline for the Diagnosis, Treatment, and Prevention of Overweight and Obesity in Adults (IMSS 46-08), over six months, with a follow-up of 18 months post-intervention.
  Interventions: Other: Conventional treatment
- Overweight workshop group (Experimental): Children between 9 to 12 years old, from the Family Medicine Unit No. 23 (IMSS, Mexico City) with a BMI Z-score 1 to 2 standard deviations above the median of the established growth patterns by age and sex, and a BMI above the 85th percentile according to WHO and CDC. Treated with a workshop based on national and international guidelines for the management of overweight and obesity, and best practices for the control and reduction of overweight and obesity in school-aged children, by the Food and Agriculture Organization (FAO). The workshop will consist of a monthly session over six months for parents and children, with a follow-up of 18 months post-intervention.
  In addition to the conventional medical treatment by their physicians, according to the Clinical Practice Guidelines.
  Interventions: Other: Playful Family Education Strategy
- Obesity conventional treatment group (Active Comparator): Children between 9 to 12 years old, from the Family Medicine Unit No. 1 and 3 (IMSS, Morelos) with a BMI Z-score 3 standard deviations above the median of the established growth patterns by age and sex, and a BMI above the 97th percentile according to WHO and CDC. Treated with conventional medical treatment by their physicians, according to the Clinical Practice Guideline for the Prevention and Diagnosis of Overweight and Obesity in Children and Adolescents (SS-025-08) and the Guideline for the Diagnosis, Treatment, and Prevention of Overweight and Obesity in Adults (IMSS 46-08), over six months, with a follow-up of 18 months post-intervention.
  Interventions: Other: Conventional treatment
- Obesity reinforcement group (Experimental): Children between 9 to 12 years old, from the Family Medicine Unit No. 23 (IMSS, Mexico City) with a BMI Z-score 3 standard deviations above the median of the established growth patterns by age and sex, and a BMI above the 97th percentile according to WHO and CDC. Treated with conventional medical treatment by their physicians, according to the Clinical Practice Guideline for the Prevention and Diagnosis of Overweight and Obesity in Children and Adolescents (SS-025-08) and the Guideline for the Diagnosis, Treatment, and Prevention of Overweight and Obesity in Adults (IMSS 46-08).
  Furthermore, in addition to the previously mentioned workshop with monthly sessions over six months for parents and children, there will be reinforcement through biweekly technological algorithms. This will be followed by an 18-month post-intervention follow-up.
  Interventions: Other: Reinforced Playful Family Education Strategy

INTERVENTIONS:
Other: Conventional treatment — Conventional medical treatment by their physicians, following the Clinical Practice Guideline for the Prevention and Diagnosis of Overweight and Obesity in Children and Adolescents (SS-025-08) and the Guideline for the Diagnosis, Treatment, and Prevention of Overweight and Obesity in Adults (IMSS 46-08), over six months, with a follow-up of 18 months post-intervention.
  Arms: Obesity conventional treatment group; Overweight conventional treatment group
Other: Playful Family Education Strategy — Workshop based on national and international guidelines for managing overweight and obesity in school-aged children, by the Food and Agriculture Organization (FAO). Monthly sessions over six months for parents and children, followed by an 18-month post-intervention follow-up.
  For parents:
  * First session focuses on raising awareness about childhood obesity through counseling and nutritional advice, promoting water consumption over sugary drinks.
  * Subsequent sessions use 'case study' technique to discuss common food and nutrition challenges.
  For children:
  * Sessions follow the 'Nutritional Guidance Intervention Guide' by the National System for Integral Family Development (DIF).
  * First session encourages healthy eating habits through activities and educational games.
  * Later sessions emphasize healthy eating patterns and physical activity.
  Arms: Overweight workshop group
Other: Reinforced Playful Family Education Strategy — The previosuly created and INDAUTOR registered workshop, will be reinforced through two-week technological algorithms, such as videogames, educational videos, and digital challenges, for the children, that they must complete through their smartphone of tablet. Followed by an 18-month post-intervention follow-up.
  Arms: Obesity reinforcement group

SUMMARY:
The goal of this non-randomized clinical controlled trial is to evaluate the impact of a playful family education strategy reinforced by the use of communication technologies in childhood obesity. The main questions to answer are:

* Does a technogical reinforced ludical family strategy might reduce overweight and childhood obesity prevalence and incidence reduction?
* Can digital reinforcement might decrease body weight, BMI, body fat mass and waist circumference in overweight or obese children?
* Does dietary habits might be improved by a technologically reinforced playful family workshop?

Researchers will compare an obesity childhood digital reinforced group to an overweight control overweight group, an overweight workshop group and a childhood obesity control group to see if technological reinforcement works to reduce and prevent childhood obesity.

DETAILED DESCRIPTION:
One of the main worldwide health problems is adult and childhood obesity, due to the complications arising from this. As World Obesity Federation (WOF) reported that in 2020, a total of 1.39 billion of adults were overweight and 0.81 billions were obese; while 260 million of children were overweight and 175 millions had obesity. Additionally, in 2022 according to the Encuesta Nacional de Salud y Nutrición (ENSANUT) 2020-2022, an 19.2% of childhood overweight prevalence was reported, and 18.1% of childhood obesity, which places our country as the second place in childhood obesity worldwide, only preceded by the USA.

Although it is well-known that the main etiological factor are the poor eating habits, promoted by the excessive consumption of sweetened beverages and ultra-processed foods. Additionally to the nutritional educational programs and guidelines, some strategies have been proposed in Mexico, in an attempt to reduce its consumption, such as the tax to soft drinks and junk food, and the front labeling of foods.

However, previous studies have demonstrated that a family program with the participation of children and parents is required, but not only by the implementation of integrative workshops, but through the reinforcement and support with the use of current technologies that have confirmed an improvement in learning processes.

So, in a pursuit of lowering childhood obesity and overweight prevalence and incidence, researchers created a non-randomized multicentric clinical trial to assess the efficacy of a technologically reinforced playful family educational workshop, on the treatment and prevention of this public health problem.

For this, a total of 196 participants will be allocated into four interventional groups:

1. Overweight children control group ( n = 49 children ) : BMI above the 85th percentile, under conventional medical treatment over six months and a 18 months post-interventional follow-up.
2. Overweight children workshop group ( n = 49 children ) : BMI above the 85th percentile, under conventional medical treatment plus a playful ludical family educational workshop, over six months and a 18 months post-interventional follow-up.
3. Childhood obesity control group ( n = 49 children) : BMI above the 97th percentile, under conventional medical treatment over six months and a 18 months post-interventional follow-up.
4. Childhood obesity digitally reinforcement group ( n = 49 children ) : BMI above the 97th percentile, under conventional medical treatment, plus a playful ludical family educational workshop and technological reinforcement, over six months and a 18 months post-interventional follow-up.

The main objective is that the overweight children workshop group achieve a normal weight or maintain in an overweight status, and those with childhood obesity and digital reinforcement become overweight or reduce body weight, fat mass and waist circumference, as secondary objectives.

Nevertheless, researchers expect the improvement of dietary habits assessed by the 24-hour Food Frequency Questionnaire (FFQ) in both interventional groups, that is the overweight workshop group and the childhood obesity digitally reinforced group.

ELIGIBILITY:
Inclusion Criteria:

* School-age children aged 9 to 12 years from the Family Medicine Unit Number 23 (IMSS, Mexico City) and the Family Medicine Units Number 1 and 3 (IMSS, Morelos).
* Children accompanied by their parents who consent to participate in the study.
* Children with a BMI equal to or greater than the 85th percentile (indicating overweight or obesity) according to CDC classification.
* Children who have agreed to participate through informed consent and assent forms.
* Families with access to Wi-Fi connection or mobile internet.
* Children with digital device (Smartphone or Tablet) access, supervised by their parents.

Exclusion Criteria:

* Children undergoing in any type of weight reduction program, whether pharmacological or non-pharmacological treatment .
* Children with a prior diagnosis of endocrinological or congenital diseases, associated with obesity, such as hypothyroidism, Prader-Willi syndrome, growth hormone deficiency, Cushing's syndrome, trisomy 21, among others.
* Children with abnormal thyroid function test results.
* Children with physical limitations, such as congenital malformations, that may prevent them from engaging in moderate to intense physical activity included in the intervention.
* Participants enrolled in another research protocol of any kind.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of childhood obesity incidence and prevalence | Baseline, 3-month and 6-month evaluation from the start of intervention, and subsequently, at 6, 12 and 18 months post-intervention.
  The prevalence of obesity will be assesed by measuring the proportion of children transitioning from obesity to overweight, according to the Centers for Disease Control and Prevention (CDC) criteria for childhood obesity. And the incidence will be determined by the proportion of overweight children who maintain their overweight status over time.

SECONDARY OUTCOMES:
Body weight | Baseline, 3-month and 6-month evaluation from the start of intervention, and subsequently, at 6, 12 and 18 months post-intervention.
  It will be measured using a Seca scale with an accuracy of 0.1 kg, following standardized international procedures.
  According to previous studies, investigators anticipate a 5% body weight baseline reduction, at the end of intervention.
Body Mass Index (BMI) | Baseline, 3-month and 6-month evaluation from the start of intervention, and subsequently, at 6, 12 and 18 months post-intervention.
  It will be assessed using body weight, and height (measured with a stadiometer with an accuracy of 0.1 cm, Weighing and Measuring Station with Frankfort line, SECA model 284), following standardized international procedures.
  Using these data, BMI (kg/m²) will be calculated and children will be classified according to their BMI percentile based on WHO and CDC charts.
  Researchers expect that children classified as overweight (BMI above the 85th percentile) will achieve a normal weight by the end of the intervention, while those classified as obese (BMI ≥ 97th percentile) will shift to the overweight category. Additionally, a reduction in BMI Z score is anticipated in both interventional and reinforced groups.
Fat Mass | Baseline, 3-month and 6-month evaluation from the start of intervention, and subsequently, at 6, 12 and 18 months post-intervention.
  It will be assessed by bioimpedance with the TANITA Iron Kids BF 689 body composition analyzer.
  After intervention investigators expect a diminishment of body fat mass percentage at the end of intervention.
Waist circumference | Baseline, 3-month and 6-month evaluation from the start of intervention, and subsequently, at 6, 12 and 18 months post-intervention.
  Measured with a Seca 201 Ergonomic Waist Circumference Measuring Tape, collocated around the stand up children body between the middle point of the anterior superior iliac spine and the costal margin, after breathing out.
  They will be classified according to the Third National Health and Nutrition Examination Survey (NHANES III) waist circumference tables for Mexican American children, and a percentile above 90 will be considered as an elevated risk.
  Investigators anticipate a reduction of waist circumference at the end of intervention in the interventional and reinforced groups.
Dietary habits | Baseline, 3-month and 6-month evaluation from the start of intervention, and subsequently, at 6, 12 and 18 months post-intervention.
  It will be assessed by a 24 hour Food Frequency Questionnaire (FFQ) to capture children's usual food and drinks consumption by querying the frequency at which a predefined food list items are consumed, including portion sizes, nutrient intake (calories, fats, proteins, carbohydrates, vitamins and minerals), eating patterns (timing, frequency, and types of meals or snacks), food diversity and diet quality.
  Investigators anticipate a reduction of consumed carbohydrates, sweetened beverages, calorie and fat intake at the end of intervention. Accompanied by an improvement of eating patterns, food diversity and diet quality according to dietary guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: José de Jesús Peralta Romero, PhD, Principal Investigator — Instituto Mexicano del Seguro Social; María Fernanda Pérez Hernández, MsC, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Unidad de Investigación Médica en Bioquímica, Unidad Médica de Alta Especialidad "Dr. Bernardo Sepúlveda", Centro Médico Nacional Siglo XXI, Instituto Mexicano del Seguro Social, Mexico City, Cuauhtémoc, Mexico

IPD SHARING:
Plan to Share IPD: No